CLINICAL TRIAL: NCT00848432
Title: Risperidone Maintenance Treatment for Relapse Prevention in Schizophrenia
Brief Title: Risperidone Maintenance Treatment in Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Professor Chuan-Yue Wang, Beijing Anding Hospital of Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2004BA720A22
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2009-02-24 (Estimated); Status verified 2009-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Risperidone; Maintenance treatment; Relapse
MeSH Terms: conditions — Schizophrenia; Recurrence | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Optimal therapeutic doses of risperidone continued for 4 weeks followed by a 50% dose reduction that was maintained for at least 11 months in clinically stable schizophrenia patients
  Interventions: Drug: risperidone
- 2 (Experimental): Optimal therapeutic doses of risperidone continued for 26 weeks followed by a 50% dose reduction for at least another 6 months in clinically stable schizophrenia patients
  Interventions: Drug: risperidone
- 3 (Experimental): Optimal therapeutic doses of risperidone continued for at least 1 year in clinically stable schizophrenia patients
  Interventions: Drug: risperidone

INTERVENTIONS:
Drug: risperidone — Patients with schizophrenia who were clinically stabilized following an acute episode were randomly assigned to a 'maintenance group' (optimal therapeutic doses continued for at least 1 year), a 4-week group (optimal therapeutic doses continued for 4 weeks followed by a 50% dose reduction that was maintained for at least 11 months) or a 26-week group (optimal therapeutic doses continued for 26 weeks followed by a 50% dose reduction for at least another 6 months)
  Other Names: Risperdal

SUMMARY:
This study set out to determine the duration of maintenance treatment with therapeutic risperidone dose in schizophrenia. In a multi-center, open label, randomized, controlled study design, patients with schizophrenia who were clinically stabilized following an acute episode were randomly assigned to a 'maintenance group' (optimal therapeutic doses continued for at least 1 year), a 4-week group (optimal therapeutic doses continued for 4 weeks followed by a 50% dose reduction that was maintained for at least 11 months) or a 26-week group (optimal therapeutic doses continued for 26 weeks followed by a 50% dose reduction for at least another 6 months).

DETAILED DESCRIPTION:
Prevention of relapse is the crucial task in the maintenance treatment of schizophrenia. This study set out to determine the duration of maintenance treatment with therapeutic risperidone dose in schizophrenia. In a multi-center, open label, randomized, controlled study design, patients with schizophrenia who were clinically stabilized following an acute episode were randomly assigned to a 'maintenance group' (optimal therapeutic doses continued for at least 1 year), a 4-week group (optimal therapeutic doses continued for 4 weeks followed by a 50% dose reduction that was maintained for at least 11 months) or a 26-week group (optimal therapeutic doses continued for 26 weeks followed by a 50% dose reduction for at least another 6 months).

ELIGIBILITY:
Inclusion Criteria:

1. in- or outpatient of either sex diagnosed with DSM-IV schizophrenia
2. having been clinically stable following an acute episode for at least 4 but less than 8 weeks, with 'clinical stability' defined as a sum score of the Brief Psychiatric Rating Scale (BPRS) of less than 36 points
3. aged between 18 and 65 years
4. receiving risperidone monotherapy titrated to optimal level in the acute phase of treatment for the psychotic episode
5. local resident, living with at least one family member after discharge
6. having satisfactory treatment adherence defined by a pill count that yielded more than 80% adherence to risperidone prescription over the past 4 weeks
7. understanding the aims of the study and having signed the consent form

Exclusion Criteria:

1. taking antidepressants, mood stabilizers, and Chinese herbal remedies concomitantly with risperidone, or having received electroconvulsive therapy (ECT), or participating in any other drug trials or interventional studies over the 4 weeks before study entry
2. having a history or ongoing experience of major chronic medical or neurological condition(s) requiring treatment that would be likely to affect psychic functions
3. past or current drug/alcohol abuse other than nicotine
4. being pregnant or having plans to become pregnant, lactating, or not practicing an effective method of birth control

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2002-12; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
relapse | at least one year

SECONDARY OUTCOMES:
psychopathology; extrapyramidal side effects and other adverse events | at least one year

CONTACTS AND LOCATIONS:
Overall Officials: Chuan-Yue Wang, MD, Principal Investigator — Beijing Anding Hospital of Capital Medical University
Locations (1):
- Beijing Anding Hospital of Capital Medical University, Beijing, China

REFERENCES:
- [Derived] Bo Q, Xing X, Li T, Mao Z, Zhou F, Wang C. Menstrual Dysfunction in Women With Schizophrenia During Risperidone Maintenance Treatment. J Clin Psychopharmacol. 2021 Mar-Apr 01;41(2):135-139. doi: 10.1097/JCP.0000000000001344. PMID 33538534
- [Derived] Bo Q, Dong F, Li X, Wang Z, Ma X, Wang C. Prolactin related symptoms during risperidone maintenance treatment: results from a prospective, multicenter study of schizophrenia. BMC Psychiatry. 2016 Nov 9;16(1):386. doi: 10.1186/s12888-016-1103-3. PMID 27829454
- [Derived] Wang CY, Xiang YT, Cai ZJ, Weng YZ, Bo QJ, Zhao JP, Liu TQ, Wang GH, Weng SM, Zhang HY, Chen DF, Tang WK, Ungvari GS; Risperidone Maintenance Treatment in Schizophrenia (RMTS) investigators. Risperidone maintenance treatment in schizophrenia: a randomized, controlled trial. Am J Psychiatry. 2010 Jun;167(6):676-85. doi: 10.1176/appi.ajp.2009.09030358. Epub 2010 Mar 15. PMID 20231321